CLINICAL TRIAL: NCT00310401
Title: The Effect of Nebulized Albuterol on Donor Oxygenation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: California Transplant Donor Network (Network); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Lorraine B. Ware, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3U01HL081332-01S1 (NIH)
Record Dates: First submitted 2006-03-01; First posted 2006-04-03 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-02

CONDITIONS: Brain Death; Organ Donor; Pulmonary Edema
Keywords: brain death; organ donor; pulmonary edema; albuterol; hypoxia; lung transplantation; infiltrates
MeSH Terms: conditions — Brain Death; Pulmonary Edema; Hypoxia | interventions — Albuterol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albuterol (Experimental): Albuterol sulfate 5 mg dissolved in normal saline administered every 4 hours by nebulization
  Interventions: Drug: Albuterol
- Saline (Placebo Comparator): Saline administered every 4 hours by nebulization
  Interventions: Drug: Albuterol; Drug: Saline

INTERVENTIONS:
Drug: Albuterol — 5 mg nebulized q4h
  Other Names: salbutamol
Drug: Saline — 1.0 cc diluted with saline in identical fashion to study drug and administered by nebulizer every 4 hours
  Other Names: placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to test the effectiveness of albuterol versus placebo with the following specific aims: a) Treatment of brain dead organ donors with albuterol will reduce pulmonary edema, improve donor oxygenation, and increase the number of lungs available for transplantation, b) Developing a blood test to predict the development of primary graft dysfunction in lung transplant recipients, and c) treating brain dead organ donors with albuterol will decrease markers of primary graft dysfunction and lead to improved lung transplant recipient outcomes and to higher rates of lungs suitable for transplantation.

DETAILED DESCRIPTION:
The donor lung utilization rate in the United States remains less than 15%, and the demand for donor lungs far exceeds the available supply. The most common reasons for failure to utilize donor lungs are donor hypoxemia and/or pulmonary infiltrates. Since pulmonary edema is a common, reversible cause of hypoxemia and infiltrates in patients with brain injury, strategies to treat pulmonary edema in organ donors should lead to improved donor oxygenation and higher rates of donor lung utilization. Inhaled beta-2 agonists increase the rate of alveolar fluid clearance and reduce pulmonary edema in both animal and human lungs. In addition, our group has recently reported that the majority of human donor lungs that are rejected for transplantation have measurable pulmonary edema and respond to beta-2 agonists with increased rates of alveolar fluid clearance. Based on this compelling scientific evidence, we propose to test the efficacy of an inhaled beta-2 agonist to increase the rate of alveolar fluid clearance and reduce pulmonary edema in brain dead organ donors with the following specific aims:

Specific Aim 1: To test the effect of aerosolized albuterol on donor oxygenation in a multicenter, randomized, double-blinded, placebo-controlled trial in 500 brain dead organ donors managed over a 2 year period by the California Transplant Donor Network (CTDN).

Hypothesis 1a: Treatment of brain dead organ donors with aerosolized albuterol will improve donor oxygenation and increase the donor lung utilization rate compared to treatment with placebo.

Hypothesis 1b: Treatment of brain dead organ donors with aerosolized albuterol will reduce the severity of pulmonary edema in procured lungs compared to treatment with placebo.

Specific Aim 2: To develop and validate a panel of biological markers that can predict and diagnose acute lung injury due to primary graft dysfunction in lung transplant recipients.

Hypothesis 2a: A panel of plasma biological markers measured in brain dead organ donors that includes markers of inflammation, coagulation, endothelial injury and lung epithelial injury will predict the development of primary graft dysfunction in the lung recipient.

Hypothesis 2b: Treatment of brain dead organ donors with inhaled beta-2 agonists will lead to reductions in levels of a panel of biological markers of inflammation, coagulation, endothelial injury, and lung epithelial injury that will be associated with increased donor lung utilization and improved recipient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Brain death
* Consent for lung donation and donor research
* Release from coroner or medical examiner

Exclusion Criteria

* Age less than 14 years

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine B Ware, M.D., Principal Investigator — Vanderbilt University Medical Center; Michael A Matthay, M.D., Principal Investigator — University of California, San Francisco; Megan Landeck, RN, BSN, APC, Principal Investigator — California Transplant Donor Network
Locations (1):
- California Transplant Donor Network, Oakland, California, United States

REFERENCES:
- [Background] Ojo AO, Heinrichs D, Emond JC, McGowan JJ, Guidinger MK, Delmonico FL, Metzger RA. Organ donation and utilization in the USA. Am J Transplant. 2004;4 Suppl 9:27-37. doi: 10.1111/j.1600-6135.2004.00396.x. PMID 15113353
- [Background] Rogers FB, Shackford SR, Trevisani GT, Davis JW, Mackersie RC, Hoyt DB. Neurogenic pulmonary edema in fatal and nonfatal head injuries. J Trauma. 1995 Nov;39(5):860-6; discussion 866-8. doi: 10.1097/00005373-199511000-00009. PMID 7474001
- [Background] Simon RP. Neurogenic pulmonary edema. Neurol Clin. 1993 May;11(2):309-23. PMID 8316188
- [Background] Matthay MA, Folkesson HG, Clerici C. Lung epithelial fluid transport and the resolution of pulmonary edema. Physiol Rev. 2002 Jul;82(3):569-600. doi: 10.1152/physrev.00003.2002. PMID 12087129
- [Background] Ware LB, Fang X, Wang Y, Sakuma T, Hall TS, Matthay MA. Selected contribution: mechanisms that may stimulate the resolution of alveolar edema in the transplanted human lung. J Appl Physiol (1985). 2002 Nov;93(5):1869-74. doi: 10.1152/japplphysiol.00252.2002. PMID 12381777
- [Background] Ware LB, Wang Y, Fang X, Warnock M, Sakuma T, Hall TS, Matthay M. Assessment of lungs rejected for transplantation and implications for donor selection. Lancet. 2002 Aug 24;360(9333):619-20. doi: 10.1016/s0140-6736(02)09774-x. PMID 12241936
- [Background] Bhorade SM, Vigneswaran W, McCabe MA, Garrity ER. Liberalization of donor criteria may expand the donor pool without adverse consequence in lung transplantation. J Heart Lung Transplant. 2000 Dec;19(12):1199-204. doi: 10.1016/s1053-2498(00)00215-1. PMID 11124490
- [Background] Sundaresan S, Semenkovich J, Ochoa L, Richardson G, Trulock EP, Cooper JD, Patterson GA. Successful outcome of lung transplantation is not compromised by the use of marginal donor lungs. J Thorac Cardiovasc Surg. 1995 Jun;109(6):1075-9; discussion 1079-80. doi: 10.1016/S0022-5223(95)70190-7. PMID 7776671
- [Background] Whiting D, Banerji A, Ross D, Levine M, Shpiner R, Lackey S, Ardehali A. Liberalization of donor criteria in lung transplantation. Am Surg. 2003 Oct;69(10):909-12. PMID 14570373
- [Background] Verghese GM, Ware LB, Matthay BA, Matthay MA. Alveolar epithelial fluid transport and the resolution of clinically severe hydrostatic pulmonary edema. J Appl Physiol (1985). 1999 Oct;87(4):1301-12. doi: 10.1152/jappl.1999.87.4.1301. PMID 10517756
- [Background] Ware LB, Matthay MA. Alveolar fluid clearance is impaired in the majority of patients with acute lung injury and the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 May;163(6):1376-83. doi: 10.1164/ajrccm.163.6.2004035. PMID 11371404
- [Background] Matthay MA, Wiener-Kronish JP. Intact epithelial barrier function is critical for the resolution of alveolar edema in humans. Am Rev Respir Dis. 1990 Dec;142(6 Pt 1):1250-7. doi: 10.1164/ajrccm/142.6_Pt_1.1250. PMID 2252240
- [Background] Ware LB, Golden JA, Finkbeiner WE, Matthay MA. Alveolar epithelial fluid transport capacity in reperfusion lung injury after lung transplantation. Am J Respir Crit Care Med. 1999 Mar;159(3):980-8. doi: 10.1164/ajrccm.159.3.9802105. PMID 10051282
- [Background] Campbell AR, Folkesson HG, Berthiaume Y, Gutkowska J, Suzuki S, Matthay MA. Alveolar epithelial fluid clearance persists in the presence of moderate left atrial hypertension in sheep. J Appl Physiol (1985). 1999 Jan;86(1):139-51. doi: 10.1152/jappl.1999.86.1.139. PMID 9887124
- [Background] Sakuma T, Okaniwa G, Nakada T, Nishimura T, Fujimura S, Matthay MA. Alveolar fluid clearance in the resected human lung. Am J Respir Crit Care Med. 1994 Aug;150(2):305-10. doi: 10.1164/ajrccm.150.2.8049807.
- [Background] Sartori C, Allemann Y, Duplain H, Lepori M, Egli M, Lipp E, Hutter D, Turini P, Hugli O, Cook S, Nicod P, Scherrer U. Salmeterol for the prevention of high-altitude pulmonary edema. N Engl J Med. 2002 May 23;346(21):1631-6. doi: 10.1056/NEJMoa013183. PMID 12023995
- [Background] Perkins GD, McAuley DF, Thickett DR, Gao F. The beta-agonist lung injury trial (BALTI): a randomized placebo-controlled clinical trial. Am J Respir Crit Care Med. 2006 Feb 1;173(3):281-7. doi: 10.1164/rccm.200508-1302OC. Epub 2005 Oct 27. PMID 16254268
- [Background] Atabai K, Ware LB, Snider ME, Koch P, Daniel B, Nuckton TJ, Matthay MA. Aerosolized beta(2)-adrenergic agonists achieve therapeutic levels in the pulmonary edema fluid of ventilated patients with acute respiratory failure. Intensive Care Med. 2002 Jun;28(6):705-11. doi: 10.1007/s00134-002-1282-x. Epub 2002 May 17. PMID 12107675
- [Background] de Perrot M, Liu M, Waddell TK, Keshavjee S. Ischemia-reperfusion-induced lung injury. Am J Respir Crit Care Med. 2003 Feb 15;167(4):490-511. doi: 10.1164/rccm.200207-670SO. PMID 12588712
- [Background] Avlonitis VS, Fisher AJ, Kirby JA, Dark JH. Pulmonary transplantation: the role of brain death in donor lung injury. Transplantation. 2003 Jun 27;75(12):1928-33. doi: 10.1097/01.TP.0000066351.87480.9E. PMID 12829889
- [Background] Christie JD, Kotloff RM, Pochettino A, Arcasoy SM, Rosengard BR, Landis JR, Kimmel SE. Clinical risk factors for primary graft failure following lung transplantation. Chest. 2003 Oct;124(4):1232-41. doi: 10.1378/chest.124.4.1232. PMID 14555551
- [Background] Thabut G, Vinatier I, Stern JB, Leseche G, Loirat P, Fournier M, Mal H. Primary graft failure following lung transplantation: predictive factors of mortality. Chest. 2002 Jun;121(6):1876-82. doi: 10.1378/chest.121.6.1876. PMID 12065352
- [Background] Christie JD, Carby M, Bag R, Corris P, Hertz M, Weill D; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part II: definition. A consensus statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2005 Oct;24(10):1454-9. doi: 10.1016/j.healun.2004.11.049. Epub 2005 Jun 4. No abstract available. PMID 16210116
- [Background] de Perrot M, Snell GI, Babcock WD, Meyers BF, Patterson G, Hodges TN, Keshavjee S. Strategies to optimize the use of currently available lung donors. J Heart Lung Transplant. 2004 Oct;23(10):1127-34. doi: 10.1016/j.healun.2003.09.010. No abstract available. PMID 15477105
- See also: Organ procurement organization participating in this study. — http://www.ctdn.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Albuterol | Saline
Started | 260 | 246
Completed | 260 | 246
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol | Saline | Total
Number analyzed (Participants) | 260 | 246 | 506
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 15 | 29
  Between 18 and 65 years | 224 | 217 | 441
  >=65 years | 22 | 14 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (16) | 42 (15) | 42 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 88 | 187
  Male | 161 | 158 | 319
Region of Enrollment [Number; unit: participants]
  United States | 260 | 246 | 506

OUTCOME MEASURES:

1. Primary Outcome: Donor Oxygenation
Description: The primary outcome was the change in oxygenation as measured by change in the PaO2/FiO2 ratio from study enrollment to organ procurement
Time Frame: Change from enrollment to organ procurement (about ~40h after enrollment)
Measure: Median (Inter-Quartile Range); unit: cmH2O
Groups:
- Albuterol: Albuterol 5 mg every 4 hour by nebulization
- Saline: Saline every 4 hours by nebulization
Arm/Group | Albuterol | Saline
Number analyzed (Participants) | 260 | 246
cmH2O | 49 [-26 to 149] | 40 [-31 to 124]
Statistical Analysis 1: Comparison: Albuterol vs Saline; Paired T Test was used to compare the change in PaO2/FiO2 ratio from enrollment to procurement between albuterol and saline treated donors; Test type: Superiority or Other; p = 0.98, Paired T Test

2. Secondary Outcome: Number of Donor Lungs Used for Transplantation
Description: Number of lungs procured and used for transplantation
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Albuterol | Saline
Number analyzed (Participants) | 260 | 246
Participants | 74 | 78

3. Secondary Outcome: Lung Compliance
Description: Static compliance of the respiratory system using plateau pressure (Pplat) measured at end-inspiration and calculated using the equation static compliance = tidal volume/(Pplat - PEEP)
Time Frame: baseline and at organ procurement (about ~40h after enrollment)
Measure: Mean (Standard Deviation); unit: ml/cmH2O
Arm/Group | Albuterol | Saline
Number analyzed (Participants) | 260 | 246
ml/cmH2O
  baseline | 48 (14) | 50 (15)
  at organ procurement (mean ~40h after enrollment) | 52 (14) | 56 (38)

4. Secondary Outcome: Pulmonary Vascular Resistance
Time Frame: 72 hours
Population: Insufficient data available to analyze this outcome
Arm/Group | Albuterol | Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Chest X-ray Findings
Description: Chest radiographs were scored using a radiographic score that scored each quadrant for extent of radiographic infiltrates on a scale of 0 to 4, then summed each quadrant for a total score from 0 (no infiltrates) to 16 (extensive infiltrates in all 4 radiographic quadrants).
Time Frame: change from enrollment to organ procurement (about ~40h after enrollment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Albuterol | Saline
Number analyzed (Participants) | 260 | 246
units on a scale
  Enrollment | 4.7 (3.3) | 4.6 (3.2)
  at organ procurement (about ~40h after enrollment) | 5.0 (3.2) | 4.4 (2.8)

ADVERSE EVENTS:
Arm/Group | Albuterol | Saline
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/246
Other Adverse Events (participants affected / at risk) | 0/260 | 0/246

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No